CLINICAL TRIAL: NCT02061397
Title: The Safety of Simvastatin (SOS) in Patients With Pulmonary Lymphangioleiomyomatosis (LAM) and With Tuberous Sclerosis Complex (TSC)
Brief Title: Safety of Simvastatin in LAM and TSC
Acronym: SOS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: The LAM Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: The SOS Trial
Record Dates: First submitted 2014-01-23; First posted 2014-02-12 (Estimated); Results first posted 2020-08-25 (Actual); Last update posted 2020-08-25 (Actual); Status verified 2020-08

CONDITIONS: Lymphangioleiomyomatosis; Tuberous Sclerosis Complex
Keywords: lymphangioleiomyomatosis (LAM); tuberous sclerosis complex (TSC); simvastatin; sirolimus; everolimus
MeSH Terms: conditions — Lymphangioleiomyomatosis; Tuberous Sclerosis | interventions — Simvastatin; Sirolimus; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- simvastatin treatment arm (Experimental): Eligible patients on sirolimus or everolimus will be assigned to receive 20 mg of simvastatin once daily for a period of two months. If tolerated, the dosage of simvastatin will be advanced to 40 mg once daily in months 3 and 4.
  Interventions: Drug: Simvastatin; Drug: Sirolimus Oral Product; Drug: Everolimus Oral Product

INTERVENTIONS:
Drug: Simvastatin — Eligible patients on sirolimus or everolimus will be assigned to receive 20 mg of simvastatin once daily for a period of two months. If tolerated, the dosage of simvastatin will be advanced to 40 mg once daily in months 3 and 4.
  Other Names: trade name Zocor
Drug: Sirolimus Oral Product — Eligible patients on sirolimus will be assigned to receive 20 mg of simvastatin once daily for a period of two months. If tolerated, the dosage of simvastatin will be advanced to 40 mg once daily in months 3 and 4.
  Other Names: Rapamune
Drug: Everolimus Oral Product — Eligible patients on everolimus will be assigned to receive 20 mg of simvastatin once daily for a period of two months. If tolerated, the dosage of simvastatin will be advanced to 40 mg once daily in months 3 and 4.
  Other Names: Afinitor

SUMMARY:
The purpose of this research study is to see if simvastatin can be taken safely in patients with either LAM or TSC, who are already being treated with everolimus or sirolimus. This is the first step in looking at simvastatin as a drug that may help patients, by impacting the growth and survival of cells that make up the lung lesions that cause problems in LAM and TSC patients. The study also seeks to learn more about how simvastatin works, when given to patients being treated with everolimus or sirolimus, and to evaluate the safety and any potential benefit to patients taking this 2-drug combination.

The primary objective of this study is to determine the safety of simvastatin in the treatment of LAM-S or LAM-TS in patients on a stable (for at least 3 months) dose of sirolimus or everolimus.

Secondary objectives include:

* To assess the effect of simvastatin on forced expiratory volume in 1 second (FEV1).
* To assess the effect of simvastatin on forced vital capacity (FVC).
* To assess the effect of simvastatin on diffusing lung capacity (DLCO).
* To assess the effect of simvastatin on vascular endothelial growth factor -D (VEGF-D) serum levels.
* To assess the effect of simvastatin with questionnaire- based assessments of dyspnea, fatigue, and quality of life (QOL).
* Assess signs of clinical benefit.

DETAILED DESCRIPTION:
After providing written informed consent, study related tests/procedures will be done to ensure eligibility for the study. If found to be eligible, the participant will be given simvastatin at a starting dose of 20 mg, to be taken each evening by mouth. If after 2 months the simvastatin 20 mg dose is tolerated, the dose of simvastatin will be increased to 40 mg each evening by mouth. Doses may be adjusted as needed, should the participant experience side effects from simvastatin. The participant's dose of everolimus or sirolimus is not expected to change, as this is a dose that has been previously tolerated. If side effects occur as a result of the combination of drugs, the dosages may be adjusted by the study physician (investigator).

ELIGIBILITY:
Inclusion Criteria:

* Female, age 18 and older with clinically definitive diagnosis (biopsy proven or compatible chest CT/MRI scan) of sporadic LAM (LAM-S) or LAM associated with TS (LAM-TS).
* Treated with a stable (at least 3 months) dose of sirolimus or everolimus
* Negative pregnancy test (women of child bearing potential) at screening.
* Women of childbearing potential must be using barrier, medically acceptable contraceptive precautions.
* Signed and dated informed consent.

Exclusion Criteria:

* Age < 18 years
* Known allergy to simvastatin or currently taking simvastatin, or therapy with a medication in the same class as simvastatin within the past 30 days.
* Allergy to sirolimus or everolimus.
* Current use of other than sirolimus or everolimus investigational drug for TSC or LAM within the past 30 days.
* Use of estrogen containing medications, including birth control pills, within the 30 days prior to enrollment.
* Treatment with drugs having known metabolic interactions with statin drugs (e.g. cytochrome P450 3A4 metabolism), including ketoconazole, itraconazole, fluconazole, erythromycin, clarithromycin, azithromycin, niacin (nicotinic acid), digoxin, warfarin, sildenafil or use of strong CYP3A4 inhibitors including gemfibrozil, cyclosporine, danazol, verapamil, diltiazem, and dronedarone. amiodarone, amlodipine, and ranolazine.
* Participation in another clinical study(ies) of an investigational treatment or drug within 30 days prior to the screening visit.
* Amiodarone; within the past 30 days.
* Significant dysfunction of liver (ALT > 2 times upper limit of normal-ULN), kidney (serum creatinine > 1.5 times ULN), or blood (leucopenia (ANC<2000), anemia, Hgb < 11 gm/dl).
* History of inflammatory muscle disease or myopathy.
* Bleeding diathesis or anticoagulant therapy.
* Uncontrolled hyperlipidemia or diabetes.
* Pregnant, breast feeding, or plan to become pregnant within the next 6 months
* Inadequate contraception (must agree to barrier method)
* History of organ transplant.
* Active on transplant list.
* Severe or uncontrolled medical conditions which would cause an unacceptable safety risk or compromise compliance with the protocol.
* Unstable seizures (recent changes in pattern or anti-epileptics).
* Mental illness or cognitive deficit precluding informed consent..
* Inability to attend scheduled clinic visits or comply with study procedures.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-03; Primary Completion 2019-12-13 (Actual); Study Completion 2019-12-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vera P Krymskaya, PhD, MBA, Principal Investigator — University of Pennsylvania; Maryl Kreider, MD, MSCE, Study Director — University of Pennsylvania; Frank McCormack, MD, Study Chair — University of Cincinnati
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Krymskaya VP. Treatment option(s) for pulmonary lymphangioleiomyomatosis: progress and current challenges. Am J Respir Cell Mol Biol. 2012 May;46(5):563-5. doi: 10.1165/rcmb.2011-0381ED. No abstract available. PMID 22550272
- [Background] Goncharova EA, Goncharov DA, Fehrenbach M, Khavin I, Ducka B, Hino O, Colby TV, Merrilees MJ, Haczku A, Albelda SM, Krymskaya VP. Prevention of alveolar destruction and airspace enlargement in a mouse model of pulmonary lymphangioleiomyomatosis (LAM). Sci Transl Med. 2012 Oct 3;4(154):154ra134. doi: 10.1126/scitranslmed.3003840. PMID 23035046
- [Background] Atochina-Vasserman EN, Goncharov DA, Volgina AV, Milavec M, James ML, Krymskaya VP. Statins in lymphangioleiomyomatosis. Simvastatin and atorvastatin induce differential effects on tuberous sclerosis complex 2-null cell growth and signaling. Am J Respir Cell Mol Biol. 2013 Nov;49(5):704-9. doi: 10.1165/rcmb.2013-0203RC. PMID 23947572
- [Result] Goncharova EA, Goncharov DA, Li H, Pimtong W, Lu S, Khavin I, Krymskaya VP. mTORC2 is required for proliferation and survival of TSC2-null cells. Mol Cell Biol. 2011 Jun;31(12):2484-98. doi: 10.1128/MCB.01061-10. Epub 2011 Apr 11. PMID 21482669

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Simvastatin Treatment Arm: Simvastatin 20 mg oral daily for 2 months; if tolerated, followed by simvastatin 40 mg oral daily for 2 months
  Simvastatin: Eligible patients will be assigned to receive 20 mg of simvastatin once daily for a period of two months. If tolerated, the dosage of simvastatin will be advanced to 40 mg once daily in months 3 and 4.
Period: Simvastatin 20 mg Oral Daily for 2 Month
Arm/Group | Single Simvastatin Treatment Arm
Started | 10
Completed | 10
Not Completed | 0
Period: Simvastatin 40 mg Oral Daily for 2 Month
Arm/Group | Single Simvastatin Treatment Arm
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Single Simvastatin Treatment Arm
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.4 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10
Rate of change in FEV1 [Mean (Standard Deviation); unit: %] — The baseline measure was lung function accessed as the forced expiratory volumes (unit ml) in 1 second (FEV1) response and was calculated as the rate of change in FEV1, which was calculated as percentage of predicted.
  % | 68.7 (23.8)

OUTCOME MEASURES:

1. Primary Outcome: Safety of Simvastatin in the Treatment of LAM-S and LAM-TS Patients
Description: Safety is a primary outcome measure which will be assessed by any major changes or deterioration in patient health.
Time Frame: 5 months
Measure: Number; unit: participants
Arm/Group | Single Simvastatin Treatment Arm
Number analyzed (Participants) | 10
participants | 0

2. Secondary Outcome: Percent Predicted FEV1
Description: Lung function will be measured by FEV1: forced expiratory volume in 1s mean and calculated as % predicted +_ SD (standard deviation).
Time Frame: 5 months
Measure: Mean (Standard Deviation); unit: percent predicted FEV1
Arm/Group | Single Simvastatin Treatment Arm
Number analyzed (Participants) | 10
percent predicted FEV1 | -2.9 (3.7)

ADVERSE EVENTS:
Time Frame: 5 months
Arm/Group | Single Simvastatin Treatment Arm
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 3/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Simvastatin Treatment Arm (N=10)
Tachycardia (Cardiac disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Peripheral adema (Blood and lymphatic system disorders) | 1 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-10-04): https://cdn.clinicaltrials.gov/large-docs/97/NCT02061397/Prot_SAP_000.pdf
  • Informed Consent Form (2016-10-04): https://cdn.clinicaltrials.gov/large-docs/97/NCT02061397/ICF_001.pdf